CLINICAL TRIAL: NCT03722524
Title: Multinational Observational Uncontrolled Open Programme "The Use of TRIple Fixed-dose COmbination in the Treatment of arteriaL Hypertension: Opportunity for Effective BP Control With cOmbined Antihypertensive Therapy"
Brief Title: The Use of TrIple Fixed-dose Combination in the Treatment of Arterial Hypertension
Acronym: TRICOLOR
Status: Completed | Type: Observational
Sponsor: Servier Russia (Industry)
Responsible Party: Sponsor
Other Study IDs: IC4-06593-057-RUS
Record Dates: First submitted 2018-10-22; First posted 2018-10-29 (Actual); Results first posted 2021-03-30 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Arterial Hypertension
MeSH Terms: conditions — Hypertension | interventions — Amlodipine; Indapamide; Calcium Channel Blockers; Diuretics; Angiotensin-Converting Enzyme Inhibitors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with arterial hypertension: The patient is included in the program if prior to the study his/her doctor decided to adjust treatment, targeted at the BP control improvement, by prescription of a triple FDC of amlodipine / indapamide / perindopril arginine. The prescription of the triple FDC of amlodipine / indapamide / perindopril arginine during the program is made by the doctor's decision according to the instructions for medical use of this FDC.
  Presumably, each doctor will include 4 patients in average. It is planned to include 1,300 patients.
  Interventions: Drug: amlodipine / indapamide / perindopril arginine FDC

INTERVENTIONS:
Drug: amlodipine / indapamide / perindopril arginine FDC — CCB / diuretic / ACE inhibitor
  Other Names: CCB / diuretic / ACE inhibitor

SUMMARY:
The use of TRIple fixed-dose COmbination in the treatment of arteriaL hypertension: opportunity for effective BP control with cOmbined antihypertensive therapy.

The main aim of this study to assess the antihypertensive effectiveness effect on the 24-hour BP profile, as well as tolerability of and compliance to the treatment with a triple FDC of amlodipine / indapamide / perindopril arginine in hypertensive patients in the real clinical practice.

Type of program: Multicenter, observational, non-controlled, open-label program.

Investigators: Cardiologists and outpatient (primary care) physicians (general practitioners).

Number of patients: 1,300 hypertensive patients.

DETAILED DESCRIPTION:
It is multicenter, observational, non-controlled, open-label program. The baseline characteristics will be analyzed in all the patients who started the treatment (intention-to-treat [ITT] population). In case of significant differences between two treatment groups, the baseline characteristics will be provided for both of them.

Changes in the SBP and DBP (with the corresponding confidence intervals) will be assessed in the patients who completed the program without major deviations from protocol (per-protocol population [PPP]).

The analysis of parameters with normal distribution will be performed using the Student's t-test for paired measurements; otherwise the non-parametric Wilcoxon test will be used. The percentage of patients with normalized BP, as well as the percentage of patients who responded to treatment (with 95% confidence intervals), will be calculated.

Questionnaires: The score for each scale will be calculated as the sum of scores for questions constituting the scale.

Assessment of the AEs will be carried out in all the patients who started the treatment (ITT population).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 79 years
* Essential hypertension
* Patient's consent to participate in the program
* Doctor's decision to prescribe FDC of amlodipine / indapamide / perindopril arginine, according to the instruction for use, prior to the inclusion in the program.

Exclusion Criteria:

* Symptomatic, or secondary arterial hypertension
* Office BP ≥ 180/110 mm Hg on treatment (at V0 visit)
* History of myocardial infarction, unstable angina, or cerebrovascular accident within the past 1 year
* CHF of class III-IV NYHA
* Type I diabetes or decompensated type 2 diabetes
* Diseases with severe organ dysfunction (hepatic failure, renal failure, etc.)
* Contraindications to or known intolerance of dihydropyridine calcium channel blockers (including amlodipine) and/or indapamide and/or ACE inhibitors (including perindopril) and/or their fixed combination
* Inability to understand the nature of the program and/or to follow the doctor's recommendations, including ones for the BP self-monitoring.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with uncontrolled arterial hypertension who needs triple antihypertensive combinations in a single tablet
Sampling Method: Non-Probability Sample
Enrollment: 1247 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2019-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natatya LOGUNOVA, Study Chair
Locations (51):
- Russia (51):
  - City Policlinic #3, Al'met'yevsk
  - City Policlinic # 9, Barnaul
  - City Policlinic # 7, Belgorod
  - City Hospital # 2, Bryansk
  - City Policlinic # 8, Chelyabinsk
  - City Policlinic # 2, Cherepovets
  - City Policlinic # 8, Irkutsk
  - City Policlinic # 5, Ivanovo
  - City Hospital # 1, Izhevsk
  - City Policlinic # 18, Kazan'
  - City Policlinic # 5, Kemerovo
  - City Policlinic # 15, Khabarovsk
  - City Policlinic # 2, Kirov
  - City Policlinic # 7, Krasnoyarsk
  - City Policlinic # 7, Kursk
  - FSBI NMIC of Cardiology of the Ministry of Health of Russia, Moscow
  - City Policlinic # 70, Moscow
  - City Policlinic # 2, Murmansk
  - City Policlinic # 17, Nizhny Novgorod
  - City Hospital # 2, Novokuznetsk
  - City Policlinic # 14, Novosibirsk
  - City Policlinic # 2, Omsk
  - Clinic PROM-MED, Orenburg
  - City Policlinic # 2, Oryol
  - Policlinic of Regional Clinic Hospital, Penza
  - Medical Center "Alfa-Center", Perm
  - City Policlinic # 4, Petrozavodsk
  - City Policlinic # 3, Pskov
  - City Policlinic # 42, Rostov-on-Don
  - City Policlinic # 2, Ryazan
  - City Policlinic # 27, Saint Petersburg
  - City Policlinic # 8, Samara
  - City Policlinic # 2, Saratov
  - City Policlinic # 2, Sevastopol’
  - Policlinic of Russian railway, Smolensk
  - City Policlinic # 2, Stary Oskol
  - City Policlinic # 3, Syktyvkar
  - City Policlinic # 6, Tambov
  - City Policlinic # 2, Tolyatti
  - City Policlinic # 2, Tomsk
  - Policlinic VIRMED, Tula
  - City Policlinic # 3, Tyumen
  - City Policlinic # 46, Ufa
  - City Policlinic # 4, Veliky Novgorod
  - City Policlinic # 4, Vladimir
  - City Policlinic # 4, Vladivostok
  - City Policlinic # 15, Volgograd
  - City Policlinic # 3, Vologda
  - City Policlinic # 7, Voronezh
  - City Policlinic # 1, Yaroslavl
  - City Policlinic # 3, Yekaterinburg

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Arterial Hypertension: The patient is included in the program if prior to the study his/her doctor decided to adjust treatment, targeted at the BP control improvement, by prescription of a triple FDC of amlodipine / indapamide / perindopril arginine. The prescription of the triple FDC of amlodipine / indapamide / perindopril arginine during the program is made by the doctor's decision according to the instructions for medical use of this FDC.
  Presumably, each doctor will include 4 patients in average. It is planned to include 1,300 patients.
  amlodipine / indapamide / perindopril arginine FDC: CCB / diuretic / ACE inhibitor
Period: Overall Study
Arm/Group | Patients With Arterial Hypertension
Started | 1247
Completed | 1148
Not Completed | 99
Not completed — Protocol Violation | 86
Not completed — Adverse Event | 7
Not completed — Lost to Follow-up | 1
Not completed — Reason is not stated | 1
Not completed — Physician Decision | 1
Not completed — Patient's decision (refusal to continue participation) | 3

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Arterial Hypertension
Number analyzed (Participants) | 1148
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 810
  >=65 years | 338
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.24 (10.48)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: No gender was indicated for 10 patients
  Participants
    number analyzed (Participants) | 1138
    Female | 687
    Male | 451
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 1148
Region of Enrollment [Number; unit: participants]
  Russia | 1148
Patients with arterial hypertension [Count of Participants; unit: Participants] | 1148

OUTCOME MEASURES:

1. Primary Outcome: The Mean Systolic BP Changes (mm Hg) at the Visit 4 vs. Baseline
Description: Changes in the mean office systolic BP levels (in mm Hg) in the sitting position Blood pressure was measured in accordance with the guidelines of the European Society of Hypertension (ESH) using the auscultatory or oscillometric method and a semi-automated sphygmomanometer. Before taking measurements, the patient remained in a sitting position for 3-5 minutes. Blood pressure was determined on each arm, and the arm with the highest value was taken as the reference. Measurements were taken thrice in the sitting position of a patient, and the average of the second and third BP measurements on the reference arm with an interval of at least 1-2 minutes was recorded.
Time Frame: Baseline, 3 months
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Patients With Arterial Hypertension
Number analyzed (Participants) | 1148
mm Hg | 33.47 (11.70)

2. Primary Outcome: The Mean Diastolic BP Changes (mm Hg) at the Visit 4 vs Baseline.
Description: Changes in the mean office diastolic BP levels (in mm Hg) in the sitting position
Time Frame: Baseline, 3 months
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Patients With Arterial Hypertension
Number analyzed (Participants) | 1148
mm Hg | 14.34 (8.63)

3. Secondary Outcome: Percentage of Patients Who Achieved the Target Office BP Levels (SBP <140 mm Hg and DBP <90 mm Hg) at Visit 4 vs Baseline
Description: The assessment of the target office BP levels (SBP <140 mm Hg and DBP <90 mm Hg) was performed in accordance with ESC Guidelines for the management of arterial hypertension (2013)
Time Frame: Baseline, 3 months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Patients With Arterial Hypertension
Number analyzed (Participants) | 1148
percentage of patients | 93.38 [91.74 to 94.72]

4. Secondary Outcome: The Mean Standardized Score of the Physical Component of the Quality of Life Questionnaire The Short Form (36) Health Survey at Visit 4 vs Baseline
Description: Change in the mean score of the of the physical component of the The Short Form (36) Health Survey (SF-36) survey.
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Time Frame: Baseline, 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients With Arterial Hypertension
Number analyzed (Participants) | 1148
score on a scale | 13.64 (18.06)

5. Secondary Outcome: The Mean Standardized Score of the Mental Component of the Quality of Life Questionnaire The Short Form (36) Health Survey at Visit 4 vs Baseline
Description: Change in the mean score of the of the physical component of the SF-36 survey Change in the mean score of the of the physical component of the The Short Form (36) Health Survey (SF-36) survey.
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Time Frame: Baseline, 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients With Arterial Hypertension
Number analyzed (Participants) | 1148
score on a scale | 23.57 (13.79)

ADVERSE EVENTS:
Time Frame: 10 months
Arm/Group | Patients With Arterial Hypertension
All-Cause Mortality (participants affected / at risk) | 0/1148
Serious Adverse Events (participants affected / at risk) | 3/1148
Other Adverse Events (participants affected / at risk) | 9/1148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Arterial Hypertension (N=1148)
tooth abscess (Immune system disorders) | 1 (1) — for which the surgical treatment was performed
exacerbation of chronic pyelonephritis (Immune system disorders) | 1 (1) — which was stopped by administration of antibiotics)
unstable angina (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Arterial Hypertension (N=1148)
arterial hypotension with BP of 80/50 mm Hg and weakness (Vascular disorders) | 1 (1)
treatment inefficacy (Vascular disorders) | 1 (1)
unstable angina (Vascular disorders) | 1 (1)
cough (Cardiac disorders) | 5 (5)
arterial hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-06-25): https://cdn.clinicaltrials.gov/large-docs/24/NCT03722524/Prot_SAP_000.pdf
  • Informed Consent Form (2018-06-25): https://cdn.clinicaltrials.gov/large-docs/24/NCT03722524/ICF_001.pdf